CLINICAL TRIAL: NCT04208750
Title: Clinical Investigation of the Vision-R800 Device. Understanding the Value of High Precision Refractions and Lenses to Optometrists and Patients. Phase 2
Brief Title: Clinical Investigation of the Vision-R800 Device.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pete Kollbaum, OD, PhD (Other)
Responsible Party: Sponsor-Investigator, Pete Kollbaum, OD, PhD, Associate Professor, Associate Dean for Research, and Director of the Borish Center for Ophthalmic Research, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Kollbaum003
Record Dates: First submitted 2019-11-14; First posted 2019-12-23 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Myopia; Hyperopia; Astigmatism; Presbyopia
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- R-Refraction (Experimental)
  Interventions: Device: Vision R-800 Phoropter; Device: Standard Phoropter
- S-Refraction (Active Comparator)
  Interventions: Device: Vision R-800 Phoropter; Device: Standard Phoropter

INTERVENTIONS:
Device: Vision R-800 Phoropter — Refraction utilizing the Vision R-800 Phoropter with resulting glasses
Device: Standard Phoropter — Refraction utilizing the standard phoropter with resulting glasses

SUMMARY:
Randomized, bilateral, cross-over dispensing study of a standard and VR800 refraction and associated spectacle lenses.

ELIGIBILITY:
Inclusion Criteria:

* current adaptated progressive addition lens wearer, if bifocal lens required
* wearable pair of glasses < 2 years old
* wear glasses at least 6 hours per day

Exclusion Criteria:

* Eye Disease with an impact on visual acuity or binocular vision abnormalities (by self-report)
* Formal training in optometry, vision science or in the eyecare field

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Clinical Optics Research Lab, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- R-Refraction Then S-Refraction; S-Refraction Then R-Refraction: Vision R-800 Phoropter: Refraction utilizing the Vision R-800 Phoropter with resulting glasses
  Standard Phoropter: Refraction utilizing the standard phoropter with resulting glasses
Period: Overall Study
Arm/Group | R-Refraction Then S-Refraction | S-Refraction Then R-Refraction
Started | 58 | 61
Visit 2 | 58 | 61
Visit 3 | 58 | 53
Visit 4 | 43 | 47
Completed | 42 | 46
Not Completed | 16 | 15
Not completed — Lost to Follow-up | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R-Refraction Then S-Refraction | S-Refraction Then R-Refraction | Total
Number analyzed (Participants) | 58 | 61 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 8 | 14
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.19 (17.57) | 38.28 (18.81) | 39.77 (18.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 11 | 18 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 52 | 60 | 112
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 48 | 47 | 95
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 61 | 119
Subject Classification [Count of Participants; unit: Participants] — young adult = someone without presbyopia, does not require a near addition presbyope = someone with presbyopia, requires a near addition
  Participants
    Count : Young Adults | 27 | 33 | 60
    Count : Presbyopes | 31 | 28 | 59
Subject Classification: Mean Age [Mean (Standard Deviation); unit: years] — young adult = someone without presbyopia, does not require a near addition presbyope = someone with presbyopia, requires a near addition Population: Sub-populations of participants were assessed for this baseline measure (young adults and presbyopes).
  years
    Young Adults: number analyzed (Participants) | 27 | 33 | 60
    Young Adults | 23.89 (7.27) | 22.06 (5.52) | 22.88 (6.38)
    Presbyopes: number analyzed (Participants) | 31 | 28 | 59
    Presbyopes | 56.26 (6.07) | 57.39 (7.06) | 56.80 (6.52)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Questionnaire Response
Description: Patient questions of refraction preference for quickness, efficiency, comfort, and stress
Time Frame: at Visit 5 (final visit), up to 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-Refraction Then S-Refraction | S-Refraction Then R-Refraction
Number analyzed (Participants) | 42 | 46
Participants
  Quickness: Prefer VR800 | 22 | 32
  Quickness: Prefer Standard | 5 | 3
  Quickness: No Preference | 15 | 11
  Efficiency: Prefer VR800 | 25 | 26
  Efficiency: Prefer Standard | 4 | 4
  Efficiency: No Preference | 13 | 16
  Comfort: Prefer VR800 | 26 | 21
  Comfort: Prefer Standard | 5 | 6
  Comfort: No Preference | 11 | 19
  Stress: Prefer VR800 | 16 | 19
  Stress: Prefer Standard | 7 | 10
  Stress: No Preference | 19 | 17
Statistical Analysis 1: Comparison: R-Refraction Then S-Refraction vs S-Refraction Then R-Refraction; Added the number of participants from each study arm who preferred each refraction type and then converted it to the proportions; Test type: Other — Difference between independent proportions; For each outcome, we compared the proportion of participants from both study arms who preferred the VR800 refraction to the proportion of participants who preferred the Standard refraction using a 2-sample test for equality of proportions

ADVERSE EVENTS:
Time Frame: 5 weeks for each participant
Arm/Group | R-Refraction | S-Refraction
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/119
Other Adverse Events (participants affected / at risk) | 0/119 | 0/119

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic this study was interrupted. Therefore, obtaining complete in-office data for some subjects was not possible. However, for all subjects possible at-home data was still obtained, as well as any in-office data that could be obtained remotely. Under allowed protocol deviation, some data was also collected in July following re-opening of the lab. We did rule out an effect of in-office as compared to remote data due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT04208750/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04208750/SAP_001.pdf